CLINICAL TRIAL: NCT07072481
Title: Sustaining Innovative Tools to Expand Youth-Friendly HIV Self-Testing
Acronym: S-ITEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Nigerian Institute of Medical Research (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202312092; UG1HD113156 (NIH)
Record Dates: First submitted 2025-06-17; First posted 2025-07-18 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: HIV/AIDS; Sexually Transmitted Diseases
Keywords: HIV Prevention; HIV self-testing; Young people
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study protocol will involve undertaking a prospective three-year assessment of the sustained intervention focused on the sustainment of the 4YBY core elements and uptake of HIV prevention services (HIV testing/retesting, STI testing/treatment, PrEP adherence), sustained capacity to implement the 4YBY program, youth engagement, and reach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard arm (4YBY-S) (Active Comparator): All Community-Based Organizations (CBOs) will implement 4YBY activities, focusing on three main components: providing HIV self-testing bundles and navigation to youth-friendly clinical sites, utilizing trained community health workers for service delivery, and facilitating peer-to-peer support among youth participants. CBOs will complete an organizational readiness survey to evaluate their capacity for implementing 4YBY.
  Interventions: Behavioral: Activities; Behavioral: Benefits; Behavioral: Capacity
- Enhanced Arm (4YBY-E) (Experimental): Cluster randomization will occur using a parallel group approach at the community level. Communities and their corresponding CBOs will be randomized 1:1 to two clusters in 40 community sites and CBOs. The 4YBY-E package will include the 4YBY-S (CBO will implement 4YBY activities, focusing on three main components: providing HIV self-testing bundles and navigation to youth-friendly clinical sites, utilizing trained community health workers for service delivery, and facilitating peer-to-peer support among youth participants) with enhanced (4YBY-E) interventions using the PLAN (People, Learning, Adaption, and Nurture) approach for sustainability and will be measured at 24 months for sustained activities, benefits, and capacity over time using both qualitative and quantitative data.
  NOTE: In this arm, the investigators will have 4YBY-S + 4YBY-E
  Interventions: Behavioral: Activities-S; Behavioral: Benefits-S; Behavioral: Capacity-S; Behavioral: People; Behavioral: Learning Meetings; Behavioral: Adaptation Monitoring; Behavioral: Nurturing Coaches

INTERVENTIONS:
Behavioral: Activities — Activities include the implementation of the three main components of 4YBY that include;
  1) provision of HIV self-testing bundles and navigation to youth-friendly clinical sites for sexually transmitted infection screening to recruited youth participants; 2) use of trained community health workers to implement the HIV self-testing bundles and STI screening services to recruited youth participants; and 3) peer-to-peer support and supervision on what works or does not work with implementing 4YBY services among recruited youth participants.
  Arms: Standard arm (4YBY-S)
Behavioral: Benefits — The benefits are conceptualized at the individual, community and CBO levels. At the individual level, at-risk youth gain access to HIV prevention services and educational materials. Community outreach will tailor educational materials to local needs, enhancing the overall impact. CBOs will form academic-community partnerships, receive training, and access resources to sustain 4YBY. A quarterly learning collaborative will also promote effective implementation.
  Arms: Standard arm (4YBY-S)
Behavioral: Capacity — Following a baseline assessment, CBOs will receive initial training on 4YBY through live videoconferences, with options for self-study for those unable to attend. Training will cover research evidence, implementation procedures, and necessary tools. Refresher training will occur every six months, ensuring ongoing support. Young people will engage in educational meetings to improve program uptake, assess quality, and enhance long-term retention.
  Arms: Standard arm (4YBY-S)
Behavioral: Activities-S — Activities include the implementation of the three main components of 4YBY that include; 1) provision of HIV self-testing bundles and navigation to youth-friendly clinical sites for sexually transmitted infection screening to recruit youth participants; 2) use of trained community health workers to implement the HIV self-testing bundles and STI screening services to recruited youth participants; and 3) peer-to-peer support and supervision on what works or does not work with implementing 4YBY services among recruited youth participants.
  Arms: Enhanced Arm (4YBY-E)
Behavioral: Benefits-S — The benefits are conceptualized at the individual, community, and CBO levels. At the individual level, at-risk youth gain access to HIV prevention services and educational materials. Community outreach will tailor educational materials to local needs, enhancing the overall impact. CBOs will form academic-community partnerships, receive training, and access resources to sustain 4YBY. A quarterly learning collaborative will also promote effective implementation.
  Arms: Enhanced Arm (4YBY-E)
Behavioral: Capacity-S — Following a baseline assessment, CBOs will receive initial training on 4YBY through live videoconference, with options for self-study for those unable to attend. Training will cover research evidence, implementation procedures, and necessary tools. Refresher training will occur every six months, ensuring ongoing support. Young people will engage in educational meetings to improve program uptake, assess quality, and enhance long-term retention.
  Arms: Enhanced Arm (4YBY-E)
Behavioral: People — Sustainability teams will be established in CBOs to lead the implementation of their sustainability blueprint for 4YBY. These teams will train staff, monitor goals, and provide feedback on performance and progress over time
  Arms: Enhanced Arm (4YBY-E)
Behavioral: Learning Meetings — CBOs will participate in bi-weekly collaborative meetings to enhance their sustainability efforts, share lessons learned, and support one another. These meetings will focus on creating a supportive learning environment and reinforcing leadership that promotes continuous learning.
  Arms: Enhanced Arm (4YBY-E)
Behavioral: Adaptation Monitoring — CBOs will adapt best practices for their sustainability plans using the FRAME-IS framework to ensure that strategies meet local needs while documenting the modifications and maintained elements over time.
  Arms: Enhanced Arm (4YBY-E)
Behavioral: Nurturing Coaches — Trained coaches will provide individualized support to CBOs, holding weekly office hours to assist with their sustainability plans, monitor progress, and address site-specific barriers to change.
  Arms: Enhanced Arm (4YBY-E)

SUMMARY:
Sustaining Innovative Tools to Expand Youth-Friendly HIV Self-Testing (S-ITEST), locally known as 4 Youth by Youth (4YBY) in Nigeria, builds on the investigator's previous efforts, which are detailed in ClinicalTrial ID#: NCT04070287, NCT03874663, and NCT04710784. Many adolescents and young adults (AYA, 14-24 years old) in Nigeria have a substantial HIV risk but do not receive adequate HIV prevention services. While pre-exposure prophylaxis (PrEP), HIV self-testing, sexually transmitted infection (STI) testing, and linkage to AYA-friendly clinical services are essential, they have not been widely implemented or sustained in Nigeria. In this study, the investigators aim to 1) use participatory approaches (i.e., crowdsourcing, designathons, and participatory learning communities (PLC)) to develop sustainability strategies that sustain 4YBY in participating community sites served by recruited community-based organizations; 2) test the effects of the standard 4YBY implementation versus standard with enhanced sustainability strategy on site-level adoption and sustainability of the 4YBY intervention across 24 months in participating community sites (n=40) and community-based organizations (n=20); and 3) characterize and estimate the impact and cost-effectiveness of sustaining 4YBY over time. Guided by youth participatory action research (YPAR), the PEN-3 cultural model, Proctor's Implementation Outcomes Framework, and the Consolidated Framework for Implementation Research (CFIR), this study intends to support community-based organizations in implementing and sustaining the 4YBY intervention to increase the uptake of HIV prevention services while optimizing resource allocation to achieve sustainability in collaboration between the Washington University School of Medicine, the University of North Carolina at Chapel Hill, Georgia State University, George Washington University, Monash University, Wake Forest University School of Medicine, and the Nigerian Institute of Medical Research (NIMR).

DETAILED DESCRIPTION:
Utilizing a participatory approach, an open call for submissions was published to engage young people in partnerships with certified community-based organizations in Nigeria. This initiative encouraged them to share their ideas, experiences, and perspectives on how community-based organizations can sustain or enhance HIV self-testing (HIVST) and youth-friendly preventive services for at-risk adolescents and young adults. During the open call, 123 submissions were received from 178 young adults and adolescents aged 14-24, offering a variety of capacity-building and adaptable ideas, such as peer health education and community engagement activities. In the designathon phase, where youth refined their ideas, 10 teams comprising 40 participants were involved, with 24 teams focusing on mobile health outreach, 8 adapting health messaging to sports, and 8 creating safe spaces for marginalized communities.

Five teams (n=20) were invited to a 4-week hybrid innovative Bootcamp to further refine their sustainment strategy, which involved training the trainers (1 team), tailoring services (1 team), creating safe spaces (1 team), modifying vans (1 team), and adapting health messaging for sporting events (1 team). All teams were awarded prizes. Strategies from all teams were combined to form the enhanced sustainability strategy for this clinical trial. In this hybrid type 2 implementation-effectiveness trial, cluster randomization will occur in a parallel group approach, with phased enrollment to standard 4YBY for all study arms, followed by an enhanced condition for CBOs randomized to the intervention condition. This study protocol will involve undertaking a prospective three-year assessment of the sustained intervention focused on the sustainment of the 4YBY core elements and uptake of HIV prevention services (HIV testing/ retesting, STI testing/treatment, PrEP adherence), sustained capacity to implement the 4YBY program, youth engagement, and reach

Step 1: Participant enrollment and baseline data collection. This will involve recruiting youth to participate in the randomized controlled trial. Participant recruitment strategies will include social media, online, event- and venue-based, participant referral, and community and school-based referrals. Participant enrollment will be completed by the study team.

Step 2: Intervention implementation. Following participant recruitment and enrollment in the study. All 40 sites will receive standard 4YBY implementation (4YBY-S), with 20 sites with matched CBOs randomized to receive standard with enhanced sustainability strategy (4YBY-E). 4YBY-S includes the continuation of standard 4YBY activities, benefits, and capacities at all participating CBOs. The Enhanced Sustainability Strategy package includes developing formal commitments and sustainability blueprint (herein referred to as PLAN) for 4YBY at randomized CBOs that includes all goals and strategies, timeframes, and milestones as well as; 1) people (i.e. identify and prepare champions known as sustainability teams); 2) learning (create a bi-weekly collaborative to improve learning, sustainability, and network weaving that promote information sharing, collaborative problem solving and shared vision/goal with sustaining 4YBY); 3) adaptation monitoring (promote and monitor adaptation to meet local needs); and 4) access to nurturing coaches (provide supportive climate and technical assistance with sustainability as well as audit and feedback)

Step 3: The investigators will conduct follow-up surveys across all 4YBY communities and CBOs and among AYA in the cohort at baseline and every six months for 24 months. Participants will use their mobile phone numbers to access the survey in person or online. Reminders will be sent via text message. The completion of the surveys will be tracked in an online database. Follow-up surveys will also be conducted to assess intervention sustainment every six months for 24 months. Additionally, every implementation encounter (i.e., initial or ongoing training, implementation of the 4YBY program, and use of sustainment strategies by the trained CHWs) will be documented in an electronic implementation dashboard maintained by the NIMR study team that will include encounter length time, time spent on 4YBY program implementation, and a checklist of implementation and sustainment strategies used.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-24
* Condomless anal or vaginal sex in the past six months Meet PrEP-eligibility criteria according to Nigerian guidelines (sex worker, MSM, person who uses drugs, partner with HIV, or sexually exposed youth, or engagement in transactional sex)
* No history of prior PrEP use
* HIV negative based on fourth-generation test
* Current resident of the recruitment city with plans to stay in city for the next 12-24 months
* Able to complete a written survey in English (the national language of Nigeria) or Pidgin English
* All participants must agree to an informed consent and provide their cell mobile number for follow-up and retention

Exclusion Criteria:

* Younger than 14 and older than 24
* Inability to comply with the study protocol
* Illness, cognitive impairment or threatening behavior with acute risk to self or others
* No informed consent
* No contact phone number
* Do not reside in any of the LGAs

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1216 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-12-24 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent sustainment of core 4YBY elements overtime (Sustained activities) | Measured at baseline, 6 months, 12 months, 18 months, and 24 months
  Sustainment of the activities will be assessed using the sustainment outcome of the Sustainment Measurement System Scale (SMSS). This includes 4-items that assess the continued operation of 4YBY including delivering it services to intended populations overtime. All youth participants as well as CHWs and CBOs will complete this assessment
Percent sustainment of core 4YBY elements overtime (Sustained benefits) | Measured at baseline, 6 months, 12 months, 18 months, and 24 months
  The investigators will use the Sustainment Measurement System Scale (SMSS) domains focused on responsiveness to community needs and values to assess 4YBY responsiveness to youth and community needs over time. At-risk youth recruited to participate as well as CHWs and CBOs will complete 7-items measuring whether the 4YBY intervention, as implemented and sustained, currently meets their needs, is consistent with the norms and values of the CBOs, fits with the values of CBOs, communities and young people, with a shared perception of project importance by all participants.
Percent sustainment of core 4YBY elements overtime (Sustained capacity) | Measured at baseline, 6 months, 12 months, 18 months, and 24 months
  The infrastructure and capacity to support the sustainment domain of the Sustainment Measurement System Scale (SMSS) will be used to assess available resources for 4YBY implementation and sustainment over time. All youth, CHWs, and CBOs will complete surveys that assess whether 4YBY is fully integrated into the operations of their communities and CBOs, as well as plans for implementing and sustaining 4YBY.

SECONDARY OUTCOMES:
People: Youth, CHW and CBO characteristics | Measured at baseline, 6 months, 12 months, 18 months, and 24 months
  The investigators will use study-created measures to capture all youth, CHW and CBOs socio-demographic profiles. The investigators will assess program reach with youth participants and assess effectiveness outcomes among youth participants randomized to 4YBY-S versus 4YBY-E. Additionally, the investigators will use the coalitions, partnerships and networks domain of the Sustainment Measurement System Scale (SMSS) to assess support for continued operation of 4YBY, perceptions of engagement, among youth, communities and CBO's overtime. The investigators will also use the implementation climate scale, an 18-item questionnaire of implementation climate in an organization that supports evidence-based intervention adoption and use with very psychometric properties (18-items; α=0.894).
Learning | Measured at baseline, 12 months, and 24 months
  The Dimension of the Learning Organization questionnaire, a psychometrically valid assessment of learning environment will be used to explore perceptions of the degree to which the atmosphere in the CBOs encouraged learning and provided opportunities for continuous learning, inquiry and dialogue, team learning, empowerment toward a collective vision, and a learning leadership with implementing and sustaining 4YBY across participating communities and CBOs. Additionally, the investigators will use the Measure of Innovation-Specific Implementation Intention (MISII) to measure individual CHWs and CBOs' intentions to implement and sustain 4YBY before and after learning. It consists of three items that each capture an aspect of intention: plans, desire, and scope, and the scale has good internal consistency (0.90).
Adaptation | Measured at baseline, 12 months, and 24 months
  CHWs and CBOs will complete a checklist from the coding manual for FRAME-IS. The checklist will be used to capture whether they have made any adaptations to 4YBY based on patient/community characteristics, such as recruitment of at-risk youth populations or access to HIV prevention services. This outcome will also be reported as frequencies (i.e., the number of CBOs who reported making adaptations per recruit participant).
Nurturing | Measured at baseline, 12 months, and 24 months
  The Implementation Citizenship Behavior Scale (ICBS) will be used to measure the extent to which CHW and CBO's exceed expectations with supporting 4YBY implementation overtime. It consists of six items divided equally across the two dimensions: (1) helping others and (2) keeping informed. Both subscales show good internal consistency in the original study (.93 and .91, respectively), as did the total scale (.93). Additionally, the Community Citizen Behavior Scale (CCB) will be adapted for use with at-risk youth participants to measure the positive behavior of AYA towards the community and CBOs with 4YBY implementation and sustainability. It includes 27 items and five five-dimensions namely, helping behavior, keeping interpersonal harmony, involving behavior, protecting behavior, and recommending behavior with Cronbach's α value that ranges from 0.841 to 0.918
Semi-structured interviews | Measured at baseline, 12 months and 24 months
  The investigators will interview a subset of youth, CHWs, and administrators of CBOs to contextualize and extend findings from the quantitative data collection. The investigators will sample from each community and CBO at baseline. At post-implementation and follow-up, a purposive sampling strategy will be utilized to ensure representation across communities and CBOs and to capture perspectives of youth, CHWs, and CBOs who experience different outcomes within each condition (e.g., 4YBY-S vs. 4YBY-E). The interviews will assess multilevel influences on 4YBY implementation and sustainability. The interview guide will be based on the tenets of the PEN-3 cultural model and the Consolidated Framework for Implementation Research.

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Iwelunmor, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Nigerian Institute of Medical Research, Yaba, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwelunmor J, Adeoti E, Gbaja-Biamila T, Nwaozuru U, Obiezu-Umeh C, Musa AZ, Xian H, Tang W, Oladele D, Airhihenbuwa CO, Rosenberg N, Conserve DF, Yates F, Ojo T, Ezechi O, Tucker JD. Factors associated with HIV self-testing and PrEP use among Nigerian youth: Baseline outcomes of a pragmatic, stepped-wedge, cluster-randomized controlled trial. Contemp Clin Trials. 2025 Jan;148:107733. doi: 10.1016/j.cct.2024.107733. Epub 2024 Nov 14. PMID 39547480
- [Background] Nathan N, Shelton RC, Laur CV, Hailemariam M, Hall A. Editorial: Sustaining the implementation of evidence-based interventions in clinical and community settings. Front Health Serv. 2023 Mar 24;3:1176023. doi: 10.3389/frhs.2023.1176023. eCollection 2023. No abstract available. PMID 37033900
- [Background] Tucker JD, Iwelunmor J, Abrams E, Donenberg G, Wilson EC, Blachman-Demner D, Laimon L, Taiwo BO, Kuhns LM, John-Stewart GC, Kohler P, Subramanian S, Ayieko J, Gbaja-Biamila T, Oladele D, Obiezu-Umeh C, Chima KP, Jalil EM, Falcao J, Ezechi OC, Kapogiannis BG. Accelerating adolescent HIV research in low-income and middle-income countries: evidence from a research consortium. AIDS. 2021 Dec 1;35(15):2503-2511. doi: 10.1097/QAD.0000000000003049. PMID 34870930
- [Background] Iwelunmor J, Tucker JD, Ezechi O, Nwaozuru U, Obiezu-Umeh C, Gbaja-Biamila T, Oladele D, Musa AZ, Airhihenbuwa CO. Sustaining HIV Research in Resource-Limited Settings Using PLAN (People, Learning, Adapting, Nurturing): Evidence from the 4 Youth by Youth Project in Nigeria. Curr HIV/AIDS Rep. 2023 Apr;20(2):111-120. doi: 10.1007/s11904-023-00652-2. Epub 2023 Mar 29. PMID 36988831